CLINICAL TRIAL: NCT05413330
Title: Combined Phacoemulsification Surgery and Intravitreal Triamcinolone Injection Versus Stand-alone Surgery in Patients With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Corticosteroid Injection Combined With Cataract Surgery in Diabetic Eyes.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UDMS-Opthal-01-2022
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Diabete Type 2; Cataract; Triamcinolone Acetonide; Intravitreal Injection
Keywords: diabetes; phacoemulsification; intravitreal; triamcinolone acetonide; diabetic retinopathy; central subfield macular thickness; CSMT; CDVA; IOP
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cataract; Diabetes Mellitus; Diabetic Retinopathy | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Prospective randomized single-blinded clinical trial
Who Masked: Participant
Masking Description: Single (Participants)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVTA group (Experimental): Patients will receive an intravitreal injection of 4 mg/0.1 mL preservative-free triamcinolone acetonide at the end of surgery.
  Interventions: Drug: Triamcinolone Acetonide
- No injection group (No Intervention): Patients will receive no additional treatment to the standard phacoemulsification surgery.

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Intravitreal injection of 4 mg/0.1 mL preservative-free triamcinolone acetonide at the end of phacoemulsification surgery will be injected at 3.5 mm inferolateral and posterior to the limbus.
  Other Names: Kenalog
  Arms: IVTA group

SUMMARY:
The investigators aim in this study to investigate the effect of intravitreal triamcinolone acetonide injection on the development of macular edema and the progression of diabetic retinopathy. Whether this injection hastens cataract surgery results or not. The investigators will categorize the participants into two groups: the case group who will receive the injection at the end of the surgery, and the control group who will have routine cataract surgery with no extra injections.

DETAILED DESCRIPTION:
Cataract and diabetic retinopathy (DR) represent two of the top five leading causes of global impaired vision and blindness according to the WHO. Higher incidence and faster cataract progression are well-established in diabetic patients, especially those with higher glycated hemoglobin values. Further, it is estimated that up to 20% of all cataract surgery is performed on diabetic patients. The investigators aim in this study to contribute to investigating the efficacy of triamcinolone acetonide injection at the end of phacoemulsification surgery in patients with type 2 diabetes in comparison with the standard phacoemulsification surgery: whether it blunts the initiation as well as the progression of diabetic macular edema and diabetic retinopathy, and improves visual outcomes. Besides, The investigators aim to evaluate the consequences and safety of the injection.

ELIGIBILITY:
Inclusion Criteria:

* ● A history of diabetes mellitus DM type II that is well-confirmed by an endocrinologist.

  * Senile cataract that is causing visual disturbance as demonstrated by clinical examination.
  * CDVA of no more than 20/ 40, finger count and hand movement vision are included. Too.
  * Diabetic retinopathy that falls in one of the following categories according to the International Clinical Diabetic Retinopathy Disease Severity Scale: No DR- mild NPDR- moderate NPDR.
  * A healthy-looking central macula, or Clinically Significant Macular Edema (CSME), or edema that is apparent on Fundus Fluorescent Angiography (FFA) or OCT, as well as a treatment-resistant diabetic macular edema in the past 24 months or microaneurysms at foveal avascular zone (FAZ) borders not amenable to laser therapy.
  * Both sexes, Age 18 years or older.
  * One eye per patient will be included.
  * The surgery will be performed by the same surgeon and the samIOL design will be used.

Exclusion Criteria:

* • A history of diabetes mellitus DM type I that is well-confirmed by an endocrinologist or no history of DM.

  * CDVA that is better than 20/40.
  * functionally monocular patient as a result of moderate to severe visual impairment in the contralateral eye, as per the definition of the International Statistical Classification of Diseases and Related Health Problems, 10th revision (6).
  * The presence of pathologies other than diabetic retinopathy and cataract that may justify visual acuity decline (e.g. corneal disease, age related macular degeneration, macular hole, etc…).
  * patients will be excluded if they had an increased risk for developing CME in the study eye because of a complication during the current or previous intraocular surgery, intraocular inflammation or uveitis, retinal vein occlusion, or macular pathology that might influence visual function, other than diabetic macular edema.
  * Patients with pseudoexfoliation syndrome, Fuchs endothelial dystrophy, or post-traumatic cataract in the study eye.
  * Diabetic retinopathy that falls in one of the following categories according to the International Clinical Diabetic Retinopathy Disease Severity Scale: severe NPDR, proliferative DR, or vitreous hemorrhage requiring pan-retinal photocoagulation or vitrectomy.
  * Patients who used topical NSAIDs, topical or systemic corticosteroids before surgery.
  * patients who received an intravitreal injection with any kind of anti-VEGF in the study eye in the previous 6 weeks, or an intraocular or periocular corticosteroid injection in the previous 3 months.
  * patients who received PRP during the past 3 months.
  * Contraindications for any of the investigated drugs, particularly patients with glaucoma, IOP of 21mm Hg or higher, previous steroid-induced IOP elevation, or ganglion cell/ RNFL complex injury on OCT image.
  * History of steroid hypersensitivity.
  * Patients who are taking steroids PO with a total dosage of more than 5 mg/ day.
  * Pregnant and breastfeeding ladies.
  * Previous surgery on the study eye.
  * systemic bleeding in the previous 3 months, major systemic surgery in the previous 3 months, or a recent or recurrent cerebrovascular accident, myocardial infarction, or thromboembolic event.

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Change in central subfield mean macular thickness as a measurement of efficacy | T0_ 1 month- T1_ 3 months- T2_ 6 months postoperatively]
  The primary endpoint is the change in central subfield mean macular thickness in the 1 mm area (central subfield macular thickness, CSMT) as compared to baseline within the first 6 months postoperatively.
Change in diabetic retinopathy grade as a measurement of efficacy | T0: 1 month- T2: 3 months- T3: 6 months postoperatively
  The primary endpoint is the change in diabetic retinopathy grade as compared to baseline within the first 6 months postoperatively.

SECONDARY OUTCOMES:
Change in corrected distance visual acuity CDVA as a measurement of efficacy | _1 week- T1_ 1 month- T2_ 3 months- T3_ 6 months postoperatively
  CDVA measurements will be taken in metres then converted to Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts (logMAR).
ntraocular pressure (IOP) as a measurement of safety | T0: 1 week- T1: 1 month- T2: 3 months- T3: 6 months postoperatively
  IOP (in mmHg) will be measured by Goldmann applanation tonometry
No. of subjects with Adverse Events as a measurement of safety | T0: 1 week- T1: 1 month-T2: 3 months- T3: 6 months postoperatively
  An adverse event (AE) is defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigational product. All adverse events reported spontaneously by the subject or observed by the principal investigator or his staff will be recorded. Endophthalmitis in particular will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SY, Yang J, Lee YC, Park YH. Effect of a single intraoperative sub-Tenon injection of triamcinolone acetonide on the progression of diabetic retinopathy and visual outcomes after cataract surgery. J Cataract Refract Surg. 2008 May;34(5):823-6. doi: 10.1016/j.jcrs.2008.01.018. PMID 18471640
- [Background] Chung J, Kim MY, Kim HS, Yoo JS, Lee YC. Effect of cataract surgery on the progression of diabetic retinopathy. J Cataract Refract Surg. 2002 Apr;28(4):626-30. doi: 10.1016/s0886-3350(01)01142-7. PMID 11955902
- [Background] Lundstrom M, Barry P, Henry Y, Rosen P, Stenevi U. Visual outcome of cataract surgery; study from the European Registry of Quality Outcomes for Cataract and Refractive Surgery. J Cataract Refract Surg. 2013 May;39(5):673-9. doi: 10.1016/j.jcrs.2012.11.026. Epub 2013 Mar 14. PMID 23499065
- [Background] Simons RWP, Wielders LHP, Nuijts RMMA, Veldhuizen CA, van den Biggelaar FJHM, Winkens B, Schouten JSAG, Dirksen CD; ESCRS PREMED Study Group. Economic evaluation of prevention of cystoid macular edema after cataract surgery in diabetic patients: ESCRS PREMED study report 6. J Cataract Refract Surg. 2022 May 1;48(5):555-563. doi: 10.1097/j.jcrs.0000000000000785. PMID 34417781
- [Background] Mittra RA, Borrillo JL, Dev S, Mieler WF, Koenig SB. Retinopathy progression and visual outcomes after phacoemulsification in patients with diabetes mellitus. Arch Ophthalmol. 2000 Jul;118(7):912-7. PMID 10900103
- [Background] Mentes J, Erakgun T, Afrashi F, Kerci G. Incidence of cystoid macular edema after uncomplicated phacoemulsification. Ophthalmologica. 2003 Nov-Dec;217(6):408-12. doi: 10.1159/000073070. PMID 14573973
- [Background] Lee R, Wong TY, Sabanayagam C. Epidemiology of diabetic retinopathy, diabetic macular edema and related vision loss. Eye Vis (Lond). 2015 Sep 30;2:17. doi: 10.1186/s40662-015-0026-2. eCollection 2015. PMID 26605370
- [Background] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Background] Eriksson U, Alm A, Bjarnhall G, Granstam E, Matsson AW. Macular edema and visual outcome following cataract surgery in patients with diabetic retinopathy and controls. Graefes Arch Clin Exp Ophthalmol. 2011 Mar;249(3):349-59. doi: 10.1007/s00417-010-1484-9. Epub 2010 Sep 9. PMID 20827486
- [Background] Wielders LHP, Schouten JSAG, Winkens B, van den Biggelaar FJHM, Veldhuizen CA, Findl O, Murta JCN, Goslings WRO, Tassignon MJ, Joosse MV, Henry YP, Rulo AHF, Guell JL, Amon M, Kohnen T, Nuijts RMMA; ESCRS PREMED Study Group. European multicenter trial of the prevention of cystoid macular edema after cataract surgery in nondiabetics: ESCRS PREMED study report 1. J Cataract Refract Surg. 2018 Apr;44(4):429-439. doi: 10.1016/j.jcrs.2018.01.029. PMID 29778106
- [Derived] Zaher Addeen S, Shaddoud I. Combined phacoemulsification surgery and intravitreal triamcinolone injection versus stand-alone surgery in patients with type 2 diabetes: a prospective randomized trial. BMC Ophthalmol. 2022 Nov 19;22(1):445. doi: 10.1186/s12886-022-02676-5. PMID 36401233